CLINICAL TRIAL: NCT01734174
Title: Left Ventricular Volume and Ejection Fraction: Validation of Real Time 3 Dimensional Transesophageal Echocardiography
Status: Withdrawn | Type: Observational
Why Stopped: Unable to obtain 3D TTE to complete study procedure.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1207012636
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: 3D Transesophageal and Transthoracic Echocardiogram
Keywords: transesophageal and transthoracic echocardiogram; thermodilution; left ventricular volume; ejection volume
MeSH Terms: interventions — Thermodilution

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac patients: Patients having elective coronary artery bypass grafting surgery, valve repair or replacement surgery, aortic repair or replacement surgery, or any combination of these surgeries will be recruited for this study to validate measurements of left ventricular volume and ejection fraction (a quantitative measure of general heart function) as assessed by 3-dimensional transesophageal echocardiography (3D TEE) as compared to 3-dimensional transthoracic echocardiography (3D TTE). Secondarily, we will also compare the 3D TEE assessment to the 2D TEE and TTE assessment, which is routinely performed simultaneously. Last, we will compare this assessment to a third method of quantification of cardiac function via a pulmonary artery catheter using thermodilution.
  Interventions: Procedure: transesophageal echocardiography (TEE); Procedure: thermodilution; Procedure: transthoracic echocardiography (TTE)

INTERVENTIONS:
Procedure: transesophageal echocardiography (TEE) — Echocardiography is an ultrasound-based imaging technique which can be performed through the esophagus (which lies behind the heart) and is performed routinely as a monitoring and diagnostic tool at different times in the course of one cardiac surgery.
Procedure: thermodilution — A catheter is positioned in the pulmonary artery and the heart function is assessed via thermodilution which involves measuring the temperature of blood when a known volume of fluid is injected through the catheter to determine how quickly blood is carried from one part of the catheter to the other.
Procedure: transthoracic echocardiography (TTE) — Echocardiography is an ultrasound-based imaging technique which can be performed through the chest wall and is performed routinely as a monitoring and diagnostic tool at different times in the course of one cardiac surgery.

SUMMARY:
Echocardiography is an ultrasound-based imaging technique which can be performed through the esophagus (which lies behind the heart) and through the chest wall; both TEE and TTE are performed routinely as a monitoring and diagnostic tool at different times in the course of one cardiac surgery. The purpose of the study is to compare these two methods of echocardiography and comparing them to the 2D TEE and TTE assessments, which are routinely performed simultaneously. The study will also compare the echocardiography data to a third technique, thermodilution, which measures cardiac function via a pulmonary artery catheter.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass grafting surgery, valve repair or replacement surgery, aortic repair or replacement surgery, or any combination of these surgeries.
* 18 years or older

Exclusion criteria for thermodilution assessment are as follows:

* Moderate to severe tricuspid regurgitation
* Contraindications to pulmonary artery catheter placement based on the American Society of Anesthesiologist's 2003 Practice Guidelines for Pulmonary Artery Catheterization.

Exclusion criteria for performance of TEE:

* Contraindications to the performance of TEE based on the Journal of the American Society of Echocardiologists' 2011 recommendations and the American Society of Anesthesiologist Guidelines for Performance of Perioperative Transesophageal Echocardiography.
* Any degree of mitral regurgitation or aortic insufficiency above trace.

Exclusion criteria for performance of TTE, both 3D and 2D:

* Qualified echocardiographer absent or unavailable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having elective coronary artery bypass grafting surgery, valve repair or replacement surgery, aortic repair or replacement surgery, or any combination of these surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
General heart function (Left ventricular volume and ejection fraction) | During cardiac surgery
  Left ventricular volume will be assessed by 3-dimensional transesophageal echocardiography (3D TEE) and compared to data from 3-dimensional transthoracic echocardiography (3D TTE). 3D measurements will be compared to the 2D TEE and TTE assessment, which is routinely performed simultaneously. Last, this assessment will be compared to a third method of quantification of cardiac function via a pulmonary artery catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Meghann Fitzgerald, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States